CLINICAL TRIAL: NCT03936452
Title: An Open, Single-center, Phase II Study of Sintilimab, Peg-aspargase Plus Anlotinib "Sandwich"With Radiotherapy in Previously Untreated Stage I-II Extranodal NK/T Cell Lymphoma
Brief Title: Combined Treatment of Sintilimab, Peg-aspargase Plus Anlotinib in NK/T Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhiming, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-048-X01
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Natural Killer/T-Cell Lymphoma, Nasal and Nasal-Type; Early Stage; Anlotinib; Peg-aspargase; Sintilimab; Phase Two; Open; Radiotherapy
MeSH Terms: interventions — sintilimab; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Sintilimab 200mg ivdrip D1 Peg-aspargase 2500U/m2 im D1 Anlotinib 12 mg po D1-14 repeat every three weeks When patients obtained an CR or PR after the second dose of the combined regimen, they woud undergo radiotherapy after the third dose of the combined regimen. Subsequently, another three cycles of the combined regimen would be administered to these patients.
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg ivdrip D1 Anlotinib 12mg po D1-14 Peg-aspargase 2500U/m2 im D1 combined with radiotherapy
  Other Names: Peg-aspargase; Anlotinib

SUMMARY:
This study aims to investigate the treatment of previously untreated stage I-II Extranodal NK/T Cell Lymphoma with sintilimab, peg-aspargase and anlotinib, "sandwich" with radiotherapy.

The primary endpoint is the complete response rate (CRR) at the end of the treatment, and the second endpoints are CRR after two cycles of the combined regimen (CRR2), overall response rate (ORR) at the end of the treatment, survival time (OS and PFS) and toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NK/T cell lymphoma;
* Male or female: ≥18 and ≤70 years old;
* Eastern Cooperative Oncology Group (ECOG) status 0-3;
* Estimated survival time > 3 months;
* No previous anti-tumor therapy including radiotherapy, chemotherapy, targeted therapy or stem cell transplantation;
* At least one evaluable or measurable lesion complying with Lugano 2014 Standard (evaluable lesion: the examination show increased uptake of lymph nodes or extranodal areas (higher than that of the liver) by 18F-Fluorodeoxyglucose/ Positron Emission Tomography (18FDG/PET) and the PET and/or Computed Tomography (CT) features coincide with lymphoma characteristics; measurable lesion: sarcoidal lesions were longer than 15 mm or extranodal lesions were longer than 10 mm, and accompanied by increased 18FDG uptake). Increased liver diffuse 18FDG uptake without measurable lesions should be excluded.
* The main organs function well, namely, the following requirements were met one week before admission: Blood routine WBC ≥ 3.5×109/L, Hb ≥ 100g/L and PLT ≥ 90×109/L; Heart and liver function were normal (total bilirubin ≤1.5×ULN, ALT and AST ≤ 2.5×ULN), renal function was normal (serum creatinine ≤1.5×upper limitation of normal (ULN)), and without abnormal coagulation function.
* Fertile patients must undergo pregnancy tests (serum or urine) within 14 days prior to study enrollment and the results are negative, and they are willing to use effective contraception during the trial;
* The imaging evaluation was Ann Arbor stage I/II.
* Voluntary participation and signed the informed consent, good compliance, with follow-up.

Exclusion Criteria:

* Patients allergic of any of drug in this regimen;
* Pregnant or lactating women
* Participated in other clinical trials within the 4 weeks prior to enrollment;
* Previous treatments with small molecule tyrosine kinase inhibitors, including familinib,sorafenib, sunitinib, regofinib, anlotinib, furquintinib, etc.
* Imaging showed tumors have involved important blood vessels (e.g. enveloping internal carotid artery/vein), or by investigators determine highly likely during the follow-up study and cause fatal hemorrhage
* History of severe hemorrhage, or any bleeding events with a severe grade of 3 or more in CTCAE 4.0 within 4 weeks prior to enrollment
* Blood pressure unable to be controlled ideally with single antihypertensive drug therapy (Systolic blood pressure > 140 mmHg, Diastolic Blood Pressure > 90 mmHg); Clinically significant cardiovascular disease (e.g. activity) including history of CVA (within 6 months), myocardial infarction (within 6 months), unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure; serious cardiac arrhythmia beyond drug control or potentially affecting experimental therapy.
* Active ulcer, intestinal perforation or intestinal obstruction;
* History of gastrointestinal perforation within 28 days prior to enrollment;
* Various factors affecting the oral administration and absorption of drugs (such as inability to swallow, after gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.);
* Abnormal coagulation or bleeding tendency (It must be satisfied that INR is under normal range without anticoagulant within 14 days prior to signing informed consent); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues; on the premise that the international standardized ratio of prothrombin time (INR) is less than 1.5, small doses of warfarin (1 mg po, qd) or aspirin (no more than 100 mg qd) are allowed for preventive purposes.
* Arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis (venous thrombosis caused by intravenous catheterization due to precancerous chemotherapy is excluded if it has been cured judged by the researchers) and pulmonary embolism.
* Renal insufficiency: routine urine tests indicate that urine protein is more than + +, or 24 hours urine protein is more than 1.0 g.
* Suffered major surgery within 28 days prior to enrollment;
* Received strong inhibitors of CYP3A4 within a week or strong inducers of CYP3A4 within 2 weeks prior to enrollment.
* Long-term non-healing wound or incomplete-healing fracture.
* Symptomatic brain metastases (confirmed or suspected);
* Severe or uncontrolled infections
* History of psychotropic drug abuse and unable to get rid of or with mental disorders;
* History of immunodeficiency, including HIV positive testing, or other acquired, congenital immunodeficiency disorders, or organ transplantation history;
* Previous and present objective evidences including history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia and severe impairment of pulmonary function.
* History of other malignancy within the last 5 years prior to enrollment, except for cured basal cell carcinoma of skin, cervix in situ carcinoma and superficial bladder cancer;Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-04-28 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Complete response rate at the end of the treatment | 12 weeks after the last dose of the regimen
  Complete response rate at the end of the treatment

SECONDARY OUTCOMES:
Adverse events | Up to one year after the start of the study
  All the adverse events of the patients related will be assessed and graded by NCI CTCAE v4.0
Progression Free Survival (PFS) | Up to three years after the start of the study
  PFS was defined as time from study registration to first disease progression or death whichever occurred first, otherwise subject data were censored at time last known disease free.
Overall Survival (OS) | Up to three years after the start of the study
  OS was defined as time from study registration to death, and otherwise censored at time last known alive.
Complete response rate after two cycles of the combined regimen | 4 weeks after the second dose of the combined regimen
  Complete response rate after two cycles of the combined regimen
Overall response rate at the end of the treatment | 12 weeks after the last dose of the combined regimen
  Overall response rate at the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Li, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No